CLINICAL TRIAL: NCT05609032
Title: Development and Pilot Testing of the Sense2Quit App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Case Western Reserve University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Professor of Disease Prevention and Health Promotion, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT7031; 1R21CA265961-01 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-11-08 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Smoking Cessation; HIV Infections
Keywords: Sense2Quit; Tobacco Use
MeSH Terms: conditions — Smoking Cessation; HIV Infections; Tobacco Use

STUDY DESIGN:
Who Masked: Participant
Masking Description: Intervention assignment will be masked to participants only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (App Arm) (Experimental): Participants randomized to the intervention arm will receive access to the Sense2Quit App (A multi-component intervention that links a smartphone app to a smartwatch to provide real-time quit reminders to curtail relapses and avoid potential triggers), standard smoking cessation counseling, and nicotine replacement therapy.
  Interventions: Behavioral: Sense2Quit App
- Control (No Intervention): Participants randomized to the control arm will receive standard smoking cessation counseling and referral to quitline.

INTERVENTIONS:
Behavioral: Sense2Quit App — Participants in the intervention arm will receive access to Sense2Quit, a smartphone app that links to a smartwatch.
  Arms: Intervention (App Arm)

SUMMARY:
This is a pilot randomized controlled trial to examine the feasibility, acceptability and preliminary efficacy of the Sense2Quit App in a sample of 60 PLWH who smoke.

DETAILED DESCRIPTION:
The estimated 40-70% of persons living with HIV (PLWH) who smoke cigarettes experience substantial tobacco-related morbidity and mortality. For PLWH, apart from achieving and maintaining a suppressed viral load, tobacco cessation is the most important health behavior they can undertake to maximize both quality of life and life expectancy. However, the currently available evidence for improving tobacco cessation among PLWH is inadequate. Few tobacco cessation interventions have been tested among PLWH, and of those which have, there is 'very low' quality evidence that they were effective in the short-term and 'moderate' quality evidence indicating similar outcomes to controls in the long-term. Thus, it is critical to develop evidence-based tobacco cessation interventions to address the complex and unique needs of PLWH. In response to this need, the investigators propose to develop a mobile intervention for PLWH who smoke building on Sense2Quit, a multi-component intervention that links a smartphone app to a smartwatch to provide real-time quit reminders to curtail relapses and avoid potential trigger. This real-time feedback is critical especially in the first few weeks of a quit attempt.

The proposed Sense2Quit intervention for PLWH who smoke cigarettes is a novel and evidence-driven intervention using mobile technology to improve tobacco cessation. This will be the first study to develop and pilot test an innovative tobacco cessation intervention for PLWH. The final product of this study will be the basis for an R01 application to conduct a large-scale efficacy study for this population.

The investigators are confident that the proposed intervention will be a high impact intervention for improving tobacco cessation among PLWH and have long-term implications for overall improvement in the public's health.

ELIGIBILITY:
Inclusion Criteria:

* PLWH confirmed through medical records or pill bottles for antiretroviral therapy (ART)medications.
* ≥ 18 years of age;
* Own an Android smartphone;
* Understand and read English;
* Not pregnant or breastfeeding (due to contraindications for Nicotine Replacement Therapy [NRT]);
* Permanent contact information;
* Smokes ≥5 cigarettes per day for the past 30 days;
* Interested in quitting smoking within 30 days;
* Blows ≥5 ppm eCO into a breath analyzer at baseline.

Exclusion Criteria:

* Use of tobacco products other than cigarettes (i.e. cigars, piped tobacco, chew, snuff)
* Planning to move within 3 months of enrollment;
* Positive history of a medical condition that precludes nicotine patch use;
* Current use of NRT or other smoking cessation medications (e.g., Chantix or Zyban);
* Current enrollment in another smoking cessation program.
* Alcohol dependence measured through the AUDIT-C
* A household member is also participating in the Sense2Quit study (due to study contamination).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schnall R, Huang MC, Brin M, Cioe PA, Liu J, Das A, Fontalvo S, Xu W. Feasibility and Acceptability of the Sense2Quit App for Improving Smoking Cessation in PWH. AIDS Behav. 2025 Jun;29(6):1920-1929. doi: 10.1007/s10461-025-04659-1. Epub 2025 Feb 25. PMID 40000581
- [Derived] Brin M, Trujillo P, Jia H, Cioe P, Huang MC, Chen H, Qian X, Xu W, Schnall R. Pilot Testing of an mHealth App for Tobacco Cessation in People Living With HIV: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Oct 19;12:e49558. doi: 10.2196/49558. PMID 37856173

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention (App Arm) | Control
Started | 30 | 30
Completed | 26 | 29
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (App Arm) | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.97 (12.05) | 58.83 (7.90) | 56.40 (10.40)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 13 | 16 | 29
  Female | 15 | 12 | 27
  Transgender Female/Transwoman/Male-to-Female | 2 | 1 | 3
  Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 8 | 9
  Not Hispanic or Latino | 29 | 22 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 24 | 24 | 48
  White | 4 | 0 | 4
  Other | 0 | 5 | 5
  Multiracial | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Education [Count of Participants; unit: Participants]
  None | 1 | 1 | 2
  Some high school, no diploma | 6 | 8 | 14
  High school diploma or equivalent | 13 | 7 | 20
  Some College | 5 | 9 | 14
  Associate degree or technical degree | 1 | 2 | 3
  Bachelor/college degree | 1 | 3 | 4
  Professional or graduate degree | 3 | 0 | 3
Annual Income [Count of Participants; unit: Participants]
  Less than $10,000 | 14 | 9 | 23
  $10,000-$19,999 | 9 | 17 | 26
  $20,000-$39,999 | 5 | 4 | 9
  $40,000-$59,999 | 1 | 0 | 1
  Don't know | 1 | 0 | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Homosexual/gay/lesbian | 12 | 10 | 22
  Heterosexual/straight | 15 | 17 | 32
  Bisexual | 2 | 3 | 5
  Asexual | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Biochemically Verified 7-day Point Prevalence Smoking/Tobacco Abstinence at 12 Weeks
Description: 7-day point prevalence abstinence is calculated as the percentage of participants who reported no smoking/tobacco use in the 7 days prior to their 12-week follow-up visits biochemically verified by exhaled Carbon Monoxide (eCO) collected at 4 and 12 weeks via breathalyzer (Micro+TM basic Smokerlyzer®). At each of the 2 follow-up timepoints, participants with eCO levels <5 parts per million (ppm) will be classified as abstinent while participants with eCO levels ≥5ppm will be classified as not abstinent.
Time Frame: 12 weeks after baseline (or quit date if later than baseline visit)
Population: 28 of the 29 control arm participants analyzed as the smokerlyzer data was not collected from one participant at the 12 week timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (App Arm) | Control
Number analyzed (Participants) | 26 | 28
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention (App Arm) | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT05609032/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT05609032/ICF_001.pdf